CLINICAL TRIAL: NCT04237272
Title: Comparison of Leading E-cigarette Product Types on Relative Reinforcement Value and Tobacco Use Patterns Among Current Smokers
Brief Title: JUUL vs. Mod E-cigarette Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Tracy Smith, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00089701; P30CA138313 (NIH)
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Smoking; Tobacco Use
MeSH Terms: conditions — Smoking; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pod System (Active Comparator): Participants assigned to this intervention will try to pod system e-cigarette in the lab and receive a pod system e-cigarette to use for a three week sampling period.
  Interventions: Other: Pod System E-cig
- Customizable Tank (Active Comparator): Participants assigned to this intervention will try to customizable tank system e-cigarette in the lab and receive a customizable tank system e-cigarette to use for a three week sampling period.
  Interventions: Other: Customizable Tank E-cig
- Control (Active Comparator): Participants assigned to this arm will not receive any e-cigarette
  Interventions: Other: Control

INTERVENTIONS:
Other: Pod System E-cig — Participants assigned to this intervention will try to pod system e-cigarette in the lab and receive a pod system e-cigarette to use for a three week sampling period.
  Arms: Pod System
Other: Customizable Tank E-cig — Participants assigned to this intervention will try to customizable tank system e-cigarette in the lab and receive a customizable tank system e-cigarette to use for a three week
  Arms: Customizable Tank
Other: Control — Participants will not receive any e-cigarette
  Arms: Control

SUMMARY:
Some smokers who try e-cigarettes transition completely from cigarettes to e-cigarettes, but others continue to use both products, or abandon e-cigarettes and return completely to cigarettes. One factor that likely impacts these tobacco use patterns is the e-cigarette device used. The majority of e-cigarettes purchased today are one of two "types:" customizable tanks or pods. These e-cigarette types differ from each other in critical ways, like nicotine delivery and sensory characteristics, that are likely to impact use by influencing the relative reinforcement value of the product. The present study will be a randomized trial investigating the impact of e-cigarette device type on reinforcement value and use among current smokers. Current smokers (n=100) will be randomly assigned to either a control group that does not receive an e-cigarette or one of two e-cigarette types: a customizable tank, or a pod. The impact of device type on relative reinforcement value will be assessed using a choice task. Participants will also take home their assigned e-cigarette for a three-week sampling period. Primary outcomes include relative reinforcement value (choices to smoke in the lab-based choice task), cigarette smoking behavior (cigarettes smoked per day during sampling), and uptake (e-cigarette puffing episodes per day during sampling).

DETAILED DESCRIPTION:
The prevalence of e-cigarettes has risen dramatically in the United States, and the impact of these products on public health remains controversial. Proponents of e-cigarettes argue that because e-cigarettes deliver lower levels of toxicants than conventional cigarettes, they may offer reduced health risks for current smokers who switch completely. However, while e-cigarettes appear to offer a path away from smoking for a subset of smokers, a large proportion of those who try e-cigarettes abandon them after a short trial period, or continue to use both products (i.e., dual use). Complete switching from cigarettes to e-cigarettes among those who try them is modest at best. Since the ultimate impact of e-cigarettes is likely dependent on their ability to curb cigarette smoking, it is important to understand the device characteristics (in addition to user characteristics: not studied here) that contribute to their uptake. One major and perhaps most visible device factor that determines uptake is the type of e-cigarette itself. The sheer volume of e-cigarette brands makes it impossible to test the impact of each brand (over 400 estimated brands). However, most e-cigarettes can be categorized into one of four broad types with distinct characteristics: cig-a-likes, tanks, customizable tanks, and pods.

There is strong evidence that cig-a-likes deliver less nicotine, are less satisfying, and are less likely to promote switching than other device types. Thus, these devices are not included in the proposed project. Tank devices have a nicotine delivery profile differs markedly from traditional cigarettes, and thus have also not been included here. The other two types, customizable tanks and pods, corner significant portions of the e-cigarette market and differ from each other in critical ways that would be expected to impact uptake, and thus constitute our primary focus. Customizable tanks deliver nicotine in a profile that more closely models the nicotine delivery of traditional cigarettes. These devices offer a high level of customization that allows users to adjust the device until they reach their desired sensory and nicotine delivery settings. However, the customization renders them relatively complicated to learn to use. Pods (e.g., JUUL) are the newest type of e-cigarette on the market. Pods utilize nicotine salts, rather than free-base nicotine, which the company claims allows them to deliver high levels of nicotine in a profile that is comparable to traditional cigarette. They offer no customization, making them easy to use. The combination of high nicotine delivery with increased usability may increase the relative reinforcement value of these products, resulting in greater uptake than other device types. There is almost no existing research that directly compares these device types against each other. The goal of this application is to provide a preliminary assessment comparing e-cigarette device types (customizable tanks, pods) in a head-to-head design.

In a between-subjects design, adult daily smokers (n=75) who are interested in trying e-cigarettes will be randomly assigned in 1:2:2 fashion to either a control group that receives no product (n=15), or to receive one of two types of e-cigarettes to sample over a three-week period: a) customizable tank, or b) pod, (n=30/group). The design is naturalistic in that participants receiving an e-cigarette will be told to use the e-cigarette as much or as little as they would like, allowing for assessment of self-determined uptake and reinforcement. Methods include both ecological assessments (electronic daily diaries) and experimental sessions (choice and purchase tasks). Biomarkers (expired carbon monoxide) will corroborate self-reported indices of use.

ELIGIBILITY:
Inclusion Criteria:

* daily smoker
* interested in using e-cigs
* have a smartphone that can receive text messages and has access to the internet or have an e-mail account they check daily (necessary for daily diary completion)
* be at least 21 years of age

Exclusion Criteria:

* additional tobacco use criteria
* additional medical criteria

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pod System | Customizable Tank | Control
Started | 13 | 12 | 6
Completed | 13 | 10 | 3
Not Completed | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pod System | Customizable Tank | Control | Total
Number analyzed (Participants) | 13 | 12 | 6 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.23 (12.85) | 46.25 (7.56) | 52 (9.59) | 45.26 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 3 | 18
  Male | 5 | 5 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 11 | 6 | 29
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 11 | 8 | 5 | 24
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 6 | 31

OUTCOME MEASURES:

1. Primary Outcome: Choices to Smoke
Description: The percentage of choices to smoke the conventional cigarette at the Week 3 visit. Participants chose between smoking a conventional cigarette, using their assigned e-cigarette, and not using any tobacco product. Participants made the choice 10 times. Outcome is calculated as = ((number of choices to smoke / 10)*100)
Time Frame: Week 3 visit
Population: 2 participants in the customizable tank group are missing for this outcome. 1 was lost to follow up after baseline. 1 was unable to finish the Week 3 visit (missing some outcomes for this visit, but not all).
Measure: Mean (Standard Deviation); unit: Percentage of Total Choices
Arm/Group | Pod System | Customizable Tank | Control
Number analyzed (Participants) | 13 | 10 | 6
Percentage of Total Choices | 26.15 (27.85) | 30 (31.27) | 38.33 (29.27)

2. Secondary Outcome: Average Cigarettes Per Day
Description: Average number of cigarettes smoked per day during Week 3 of sampling
Time Frame: Week 3
Population: 1 person was lost to follow up after baseline in the customizable tank group.
Measure: Mean (Standard Deviation); unit: Cigarettes per Day
Arm/Group | Pod System | Customizable Tank | Control
Number analyzed (Participants) | 13 | 11 | 6
Cigarettes per Day | 10.33 (7.72) | 9.90 (7.52) | 13.99 (6.67)

ADVERSE EVENTS:
Time Frame: 3 Weeks
Description: Questionnaire at each visit asking about risks listed in the consent form as well as soliciting other adverse events that were not specifically named.
Arm/Group | Pod System | Customizable Tank | Control
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 4/13 | 9/12 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pod System (N=13) | Customizable Tank (N=12) | Control (N=6)
Burning in the Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1)
Increased Phlegm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0)
Stomachache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Throat and Mouth Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT04237272/Prot_SAP_000.pdf